CLINICAL TRIAL: NCT05475938
Title: Application of Painting Analysis and Psychotherapy in the Nursing of Children Bone Tumor
Brief Title: Application of Painting Analysis and Psychotherapy in Children With Bone Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Liuxin, Principal Investigator, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHGJ20200165
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Bone Tumors
MeSH Terms: conditions — Bone Neoplasms | interventions — Psychoanalysis

STUDY DESIGN:
Intervention Model Description: The experimental group underwent psychological evaluation, drawing analysis and psychotherapy intervention before and after chemotherapy and surgery, while the control group only underwent psychological evaluation without drawing analysis and psychotherapy intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analysis of painting (Experimental): Pathologically confirmed children with malignant bone tumors, painting therapists to explain the requirements and purpose of painting. After the patient completes the painting, the therapist makes a targeted and individualized analysis and provides psychological counseling by reflecting the patient's psychological state through painting.
  Interventions: Other: Painting therapy and psychoanalysis
- Psychological treatment (Experimental): After the patient completes the painting, the therapist makes a targeted and individualized analysis and provides psychological counseling by reflecting the patient's psychological state through painting.
  Interventions: Other: Painting therapy and psychoanalysis

INTERVENTIONS:
Other: Painting therapy and psychoanalysis — Pathologically confirmed children with malignant bone tumors, painting therapists to explain the requirements and purpose of painting. After the patient completes the painting, the therapist makes a targeted and individualized analysis and provides psychological counseling by reflecting the patient's psychological state through painting.

SUMMARY:
In the population suffering from cancer, children and teenagers are in the majority. For children with rapid development of body and mind, with the change of cognitive ability, they will feel anxiety and fear about the expected potential negative events. Painting art therapy is a kind of non-verbal psychological therapy through the interaction between the painter, the painting work and the therapist, with the painting creation activity as the intermediary. The purpose is to develop symbolic language, touch the inner subconscious, and integrate into the personality, so as to produce cognitive and behavioral changes. Painting therapy and psychological analysis can improve the treatment compliance of children bone tumor patients, make psychological nursing and health education of patients more targeted, and promote the cooperation between medical care and patients.

DETAILED DESCRIPTION:
In the population suffering from cancer, children and teenagers are in the majority. For children with rapid development of body and mind, with the change of cognitive ability, they will feel anxiety and fear about the expected potential negative events. Painting art therapy is a kind of non-verbal psychological therapy through the interaction between the painter, the painting work and the therapist, with the painting creation activity as the intermediary. The purpose is to develop symbolic language, touch the inner subconscious, and integrate into the personality, so as to produce cognitive and behavioral changes. Painting therapy and psychological analysis can improve the treatment compliance of children bone tumor patients, make psychological nursing and health education of patients more targeted, and promote the cooperation between medical care and patients. Forty pediatric bone tumor patients meeting the requirements were selected from the bone and soft tissue ward of our hospital. Twenty subjects were randomly divided into experimental group and control group. The experimental group underwent psychological evaluation, drawing analysis and psychotherapy intervention before and after chemotherapy and surgery, while the control group only underwent psychological evaluation without drawing analysis and psychotherapy intervention. This experiment was designed to evaluate the change of psychological state of children after intervention. To verify whether the intervention has improved the psychological and cognitive aspects of the children.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 7-16
2. No gender limitation
3. Pathologically confirmed patients with osteosarcoma and Ewing's sarcoma
4. Have painting ability

Exclusion Criteria:

1. Those who do not cooperate
2. Family members or patients reject this treatment technique
3. The patient has severe intellectual disability;
4. The patient's condition is in critical stage or bone marrow suppression stage or complicated with serious complications.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Psychological distress thermometer | Up to approximately 2months
  The significance of psychological distress is identified according to the score
Anxiety Screening Form for Children (SCARED) | Up to approximately 2months
  It consists of 41 items and 5 factors (somatization/panic, generalized anxiety, dissociative anxiety, social phobia and school phobia). The scale is divided into 3 levels (0 points: none; 1 mark: Sometimes. 2 marks: quite often. SCARED score ≥23 is positive, that is, the presence of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No